CLINICAL TRIAL: NCT03660085
Title: Randomized Clinical Trial of an Early vs Late Patient Empowerment Program for Men Undergoing Curative Treatment for Prostate Cancer
Brief Title: Prostate Cancer - Patient Empowerment Program
Acronym: PC-PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Gabriela Ilie, Faculty/Assistant Professor, Nova Scotia Health Authority
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PCaPRO_Halifax_001; PCaPRO_Halifax_002 (Other: NSHA)
Record Dates: First submitted 2018-08-29; First posted 2018-09-06 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical Prostatectomy; Urological Symptoms; Radiation Therapy; Mental Health; Pre-Habilitation; Exercise; Pelvic floor exercises; Intimacy and Connection; Social connection; Meditation; Stress reduction
MeSH Terms: conditions — Prostatic Neoplasms; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants receive one of two (or more) alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Early Intervention (Experimental): For 180 days participants in this arm will be exposed to the intervention and 180 days afterwards they will be exposed to the standard of care.
  Interventions: Behavioral: PC-PEP
- Arm B - Late Intervention (Active Comparator): For 180 days participants in this arm will be exposed to the standard of care and 180 days afterwards they will be exposed to the intervention.
  Interventions: Behavioral: PC-PEP

INTERVENTIONS:
Behavioral: PC-PEP — The 6 months "at home" program focuses on aerobic and strength training, pelvic floor muscle exercises, meditation, social connection, and overall healthy lifestyle practices supported with daily text message/email reminders. The aerobic (5 times/week) and strength (2 times/week) program will comprise of a single 30-minute session daily and will be individualized to each participant. Pelvic floor muscle training will include three, 10-minute sessions and mediation for 10 minutes daily. Intimacy and Connection component of PC-PEP consists of engaging in at least one form of intimacy practice prescribed, per day. Social connection will be fostered by pairing participants up with peers from the study. To encourage program compliance, study participants will receive 3 daily reminders to do their pelvic floor muscle exercises per day plus an additional motivational email daily containing helpful tips.

SUMMARY:
Each year over 20,000 men are diagnosed with prostate cancer in Canada with the majority undergoing some form of treatment option. Radical prostatectomy and/or radiation therapy are common procedures that are effective in the treatment of prostate cancer. However, they typically incur both short- and long-term side effects (e.g. urinary incontinence, sexual dysfunction, reduced physical function, etc) that can negatively impact one's quality of life. This study aims to educate and teach pre- (as opposed to most common post-) habilitation - preventive life habits aimed to empower men and address many of the issues faced by men undergoing radical prostatectomy or other active forms of prostate cancer treatments. The investigators hypothesize that daily text and email reminders, in addition to connecting men with other men undergoing similar challenges, will improve participant adherence to the pre-habilitation program. Secondary objectives will assess change in mental health, physical fitness, urological symptoms, state of relaxation, and quality of life parameters before and after the program.

DETAILED DESCRIPTION:
In a survey study of almost 400 survivors of prostate cancer (PC), we found that 17% of them suffered currently from mental health issues, and most were not on medication to address this issue. Compounding issues included urinary and sexual disfunction, poor attendance to support groups, intimacy, problems sleeping and other health problems. To address these many issues directly, with the endorsement of physicians and patients attending our regional PC integrative care conference (April 2018) and expanding on pre-habitation (pre-surgery) science, we created a Patient Empowerment Program (PEP) to be delivered from day one of diagnosis, to educate and teach the men and partners life skills/habits which are aimed to improve their fitness levels and quality of life, and to decrease treatment related side effects. This program is in line with the Auditor General of Nova Scotia's 2017 report endorsing the use of bottom-up evidence-based interventions, created from actively engaging patients in development and process. We aim to trial PC-PEP for men undergoing curative treatment for PC versus a control group receiving standard care. The PC-PEP program includes in-person and multimedia informational, physical activity, pelvic floor, stress reduction, and relationship/connection training. The men are connected with other participants to increase social support and maximize compliance. We use technology to deliver daily alerts to patients to remind them to engage in the program. A PC-PEP feasibility study of 30 men, over 28 days, showed that the program is feasible, leads to positive outcomes in patients and is highly (9.79/10) endorsed by patients. We propose a Randomized Clinical Trial assessing PC-PEP over 6 months from day one of diagnosis. We predict that PC-PEP will improve mental health (primary outcome) and other quality of life outcomes of patients compared with 'usual care'.

This is a randomized, wait-list controlled clinical trial for men newly diagnosed with PC and undergoing curative surgery and/or radiotherapy. The PEP group will receive the intervention for six months (early intervention) while the wait-list group will start the same program at the end of this intervention (late intervention; for six months). Outcomes will be assessed at baseline, six and twelve months. The primary outcome is mental health measured by the Kessler Psychological Distress Scale (K10 questionnaire) at the end of the intervention period. Multiple secondary endpoints include urinary, bowel and sexual function, fitness levels, fatigue, sleep, intimacy/sexuality concerns, relationship satisfaction, social support and surrogates of medical costs (e.g., number of visits to medical professionals).

Introducing a comprehensive empowerment program from day 1 of diagnosis may mitigate against the high levels of mental distress short and long-term suffered by hundreds of Nova Scotian men undergoing curative PC treatment every year, and the burden treatment related side effects will place on our health care system. Given that the study has the endorsement of patients, clinicians and administrators at NSHA, if proven successful it will have the evidence base needed to change the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* History of prostate cancer diagnosis
* Non-metastatic stage at start of study
* Approval from screening physician to participant in study
* Existing (or willingness to create) email account
* Ability to access and use daily email +/- text messages
* Ability to understand and speak English language
* Ability to participate in low to moderate levels of physical activity
* Scheduled for a Radical Prostatectomy (RP) or curative intent Radiotherapy (RT)(external bean or bratty) or adjuvant or salvage RT post RP. Patient on Hormone therapy are eligible if they are scheduled to undergo RP or RT.
* If deemed necessary by study physician, approval from family physician or oncologist to participate in the study

Exclusion Criteria:

* Unable to travel to Halifax for study visits (3 in total)
* Unable to access the internet and lack of a computer/cellphone to receive emails required for study intervention
* Patients being treated with Hormone therapy only
* Patients on Active Surveillance
* Patients deemed unfit to participate in low level exercise

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Mental Health | 12 months
  Kessler 10 - assessment of psychological distress pre (day 0) and post (6 months) intervention and end of study (12 months). Measured through on-line survey.

SECONDARY OUTCOMES:
General Health (Physical and Mental) Quality of Life | 12 months
  The Short Form (SF-12) Health Survey will be used to assess views about general health (physical and mental) quality of life. Change score will be calculated by taking the difference between measures taken at baseline (day 0) and post intervention (day 180).Assessment of these measures will also be completed at the end of the study (day 360). Assessed via on-line survey.
Functional, emotional and social well being | 12 month
  The Functional Assessment of Cancer Therapy-Prostate (FACT-P) will be used to measure psychosocial factors. Changes will be calculated by taking the difference between measures taken at baseline (day 0) and post intervention (day 180).Assessment of these measures will also be completed at the end of the study (day 360). Assessed via on-line survey.
Urinary, bowel, hormonal, & sexual function | 12 month
  The Expanded Prostate Index Composite (EPIC) (urinary, bowel, hormonal and sexual) and I-PSS (urinary) will be used to measure urinary function pre and post intervention. Change score will be calculated by taking the difference between measures taken at baseline (day 0) and post intervention (day 180). This will be assessed via on-line survey. Assessment of these measures will also be completed at the end of the study (day 360).
EEG (Brainwaves) | 12 month
  Electroencephalography (EEG) assessment of stress state will be measured using the Muse (IntraXon, Inc. Toronto, Ontario, Canada) neurofeedback device. Averages in relaxation brainwaves activity measurements (e.g. alpha, beta, delta, theta, and gamma) will be taken over listening to 10 minutes of relaxation music and instructions. The difference between scores at baseline (day 0) and post intervention (day 180) will be assessed. Assessment of these measures will also be completed at the end of the study (day 360). Assessment will be performed during study visits.
Heart rate variability | 12 months
  Heart rate variability (HRV) will be assessed through a HRV monitor produced by HeartMath institute. participants will be given home the device for biofeedback purposes with regards to practicing the meditation training received. The device produces scores of HRV and those at pre- (day 0) will be compared to scores at post intervention (day 180), and also at the end of the study (day 360). This will be assessed via on-line survey.
Relationship Satisfaction | 12 months
  Dyadic Assessment Scale will be used to assess relationship satisfaction at pre- (day 0) will be compared to scores at post intervention (day 180), and also at the end of the study (day 360).
Diet | 12 months
  Starting the conversation diet questionnaire will be used (developed by CHPDP). It will be assessed on-line via a survey (day 0, day 180 and day 360)
Health care utilization | 12 months
  This will be assessed online through two questions assessing number of visits to see a health care practitioner, and hospital admissions one year prior to the study and then during the year when the study was conducted.
Physical fitness: Six-minute walk test | 12 months
  Pre and post intervention assessment of physical fitness assessed to see how many meters the p[participant can walk during a timed six-minute walk test. Pre and Post scores will be taken at baseline (day 0 - pre) and post intervention (day 180 post). Assessment of these measures will also be completed at the end of the study (day 360) during study visits. Differences between the assessments will be assessed to see if the intervention had an effect.
Physical fitness: One-legged stance test | 12 months
  The length of time (in seconds) of static postural and balance control will be assessed at pre and post intervention, measured in minutes. Change score will be calculated by taking the difference between each of the pre and post measures taken at baseline (day 0) and post intervention (day 180). Assessment of these measures will also be completed at the end of the study (day 360) during study visits. Differences between the assessments will be assessed to see if the intervention had an effect.
Physical fitness: Timed sit-to-stand test | 12 months
  Pre and post intervention participants will be timed for 30 seconds to measure the amount of time they can go from sitting to standing in the allocated 30 seconds. The test will be used to test for lower limb strength. Change score will be calculated by taking the difference between each of the measures taken at baseline (day 0) and post intervention (day 180). Assessment of these measures will also be completed at the end of the study (day 360) during study visits.Differences between the assessments will be assessed to see if the intervention had an effect.
Physical fitness: Flexibility of shoulder and hamstring | 12 months
  Flexibility of shoulder and hamstring will be assessed recording the distance (in cm) rather than the degrees of the reach. Change score will be calculated by taking the difference between each of the measures taken at baseline (day 0) and post intervention (day 180). Assessment of these measures will also be completed at the end of the study (day 360) during study visits.Differences between the assessments will be assessed to see if the intervention had an effect.
Physical fitness: Grip strength | 12 months
  Pre and Post measurements of grip strength using a dynamometer will be used to test the strength of the arm and and hand forearm muscles. Change score will be calculated by taking the difference between each of the measures taken at baseline (day 0) and post intervention (day 180). Assessment of these measures will also be completed at the end of the study (day 360) during study visits.Differences between the assessments will be assessed to see if the intervention had an effect.
Height | Day one of the study
  The height of the individual will be measured in cm at the start of the program.
Weight | 12 months
  The weight of the individual participants will be measured in kg using a manual scale, in kg, at pre and post intervention. Change score will be calculated by taking the difference between each of the measures taken at baseline (day 0) and post intervention (day 180). Assessment of these measures will also be completed at the end of the study (day 360) during study visits.Differences between the assessments will be assessed to see if the intervention had an effect.
BMI - body mass index | 12 months
  Body mass index will be calculated at pre and post intervention using the height and weight scores obtained. The BMI formula we will use is: Kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared. Change score will be calculated by taking the difference between each of the measures taken at baseline (day 0) and post intervention (day 180). Assessment of these measures will also be completed at the end of the study (day 360) during study visits. Differences between the assessments will be assessed to see if the intervention had an effect.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Ilie, PhD, Principal Investigator — Nova Scotia Health Authority; Rob Rutledge, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burgher C, Ilie G, Mason R, Rendon R, Kokorovic A, Bailly G, Patil N, Bowes D, Wilke D, MacDonald C, Tsirigotis M, Butler C, Bell D, Spooner J, Rutledge RDH. Assessing the Impact of the Prostate Cancer Patient Empowerment Program (PC-PEP) on Relationship Satisfaction, Quality of Life, and Support Group Participation: A Randomized Clinical Trial. Curr Oncol. 2024 Oct 21;31(10):6445-6474. doi: 10.3390/curroncol31100479. PMID 39451783